Evaluation of Factors Associated with Patient Satisfaction and Mood-State in Regional

**Anesthesia** 

Vildan Tosuner Akpinar MD<sup>1,2</sup>, Lale Van Koroglu MD<sup>1</sup>, Hande Gurbuz Aytuluk MD<sup>1,3</sup>

1: Izmir Ataturk Training and Research Hospital; Department of Anesthesiology and

Reanimation

2: New affiliation: Izmir Bozyaka Training and Research Hospital; Department of

Anesthesiology and Reanimation

3: New affiliation: Kocaeli Derince Training and Research Hospital; Department of

Anesthesiology and Reanimation

**Trial registration:** NCT03476278

Date of the document:

Initial Release: March 17<sup>th</sup>, 2018

Study Start (Actual): January 1st, 2010

**Study Completion (Actual):** January 1<sup>st</sup>, 2011

Last Update: February 17<sup>th</sup>, 2019

**Objectives:** To evaluate factors associated with patient satisfaction from regional anesthesia procedure and mood-state of patients who underwent surgery under regional anesthesia.

**Design and Subjects:** This study was held on 300 patients who underwent surgery under regional anesthesia in Izmir Ataturk Research and Training Hospital.

**Methods:** Data collection included patient characteristics, previous anesthetic and surgical experiences, type of surgery, perioperative critical events, and preoperative information about the anesthetic procedure. Hypotension, bradycardia, pain, nausea and vomiting were rated on an ordinal scale and dichotomized as "1" for presence and "0" for absence of any of these adverse events. At the recovery room, patients were handed a questionnaire about regional anesthesia to determine patient satisfaction and mood-state during the procedure. Patients were only able to mark one option: satisfied or dissatisfied. At the same time, they were able to mark more than one option in the part of the questionnaire about mood-state: safe, unsafe, comfortable, exited, anxious. If patient was heavily sedated and too confused to participate, the questionnaire was handed at the ward after recovery.

All patients had preanesthetic evaluation prior to the surgery. The decision of general or regional anesthesia was left to the patient's primary physician anesthesiologist. Heart rate, blood pressure, and oxygen saturation were recorded every 5 minutes during the operation, and every 15 minutes at the recovery room. Complications (bradycardia, hypotension, pain, nausea and vomiting) were recorded. Patients that are clinically significant psychiatrically ill, illiterate, and patients who received general anesthesia and patients that have speech, hearing, or understanding problems were excluded from the study.

**Statistical analysis:** Data were evaluated using SPSS 16.0 (Statistical Program for Social Sciences, Chicago, II, U.S). Associations of categorical variables with patient satisfaction and

dissatisfaction were assessed using chi-square or Fisher's Exact tests. Significance of continuous variables were assessed with t-test and Mann Whitney U test. P value of <0.05 was used for statistically significance.

**Ethical Consideration:** This study was approved by the Izmir Ataturk Training and Research Hospital Institutional Review Board (Decree #32, August 10<sup>th</sup>, 2010) and written informed consent was obtained from all subjects participating in the trial. All procedures followed were in accordance with the ethical standards of the responsible committee on human experimentation and with the Helsinki Declaration of the World Medical Association.